CLINICAL TRIAL: NCT06134648
Title: A Phase I/IIa, Randomized, Observer-blind Placebo-controlled Multi-arm Study to Evaluate the Safety and Immunogenicity of an RSV/hMPV Vaccine, in Adult Participants Aged 60 Years and Older
Brief Title: Study of a Respiratory Syncytial Virus/Human Metapneumovirus Vaccine Candidate
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VBD00003; U1111-1287-8547 (Registry Identifier: ICTRP)
Record Dates: First submitted 2023-11-07; First posted 2023-11-18 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Respiratory Syncytial Virus Infection; Healthy Volunteers; Human Metapneumovirus
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Intervention Model Description: Dose-escalation (Phase I, sentinel cohort), parallel (Phase IIa, main cohort), multi-center
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sentinel, Main, and Booster Cohorts: observer-blind; for safety evaluation purposes, the Sponsor will be unblinded
  * Investigators, laboratory personnel, and participants will be blinded
  * Sponsor study staff and study staff preparing/administering the study interventions will be unblinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Sentinel Cohort: RSV/hMPV Group 0 (Dose L) (Experimental): Participants will be randomized to receive a single IM injection of RSV/hMPV vaccine candidate
  Interventions: Biological: RSV/hMPV vaccine candidate Dose L
- Sentinel Cohort: RSV/hMPV Group 1 (Dose A) (Experimental): Participants will be randomized to receive a single IM injection of RSV/hMPV vaccine candidate
  Interventions: Biological: RSV/hMPV vaccine candidate Dose A
- Sentinel Cohort: RSV/hMPV Group 2 (Dose B) (Experimental): Participants will be randomized to receive a single IM injection of RSV/hMPV vaccine candidate
  Interventions: Biological: RSV/hMPV vaccine candidate Dose B
- Sentinel Cohort: Placebo-Group 3 (Placebo Comparator): Participants will be randomized to receive a single IM injection of placebo
  Interventions: Biological: Placebo
- Main Cohort: RSV/hMPV Group 1 (Dose A) (Experimental): Participants will be randomized to receive a single IM injection of RSV/hMPV vaccine candidate
  Interventions: Biological: RSV/hMPV vaccine candidate Dose A
- Main Cohort: RSV/hMPV Group 2 (Dose B) (Experimental): Participants will be randomized to receive a single IM injection of RSV/hMPV vaccine candidate
  Interventions: Biological: RSV/hMPV vaccine candidate Dose B
- Main Cohort: Placebo-Group 3 (Placebo Comparator): Participants will be randomized to receive a single IM injection of placebo
  Interventions: Biological: Placebo
- Booster Cohort-RSV/hMPV (Experimental): Participants will be randomized to receive a determined dose of single IM injection of RSV/hMPV vaccine candidate from a subset of Main cohort
  Interventions: Biological: RSV/hMPV vaccine candidate Dose A; Biological: RSV/hMPV vaccine candidate Dose B
- Booster Cohort-Placebo (Placebo Comparator): Participants will be randomized to receive of single IM injection of placebo from a subset of Main cohort
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: RSV/hMPV vaccine candidate Dose L — Pharmaceutical form:Suspension for injection-Route of administration:Intramuscular Injection
  Arms: Sentinel Cohort: RSV/hMPV Group 0 (Dose L)
Biological: RSV/hMPV vaccine candidate Dose A — Pharmaceutical form:Suspension for injection-Route of administration:Intramuscular Injection
  Arms: Booster Cohort-RSV/hMPV; Main Cohort: RSV/hMPV Group 1 (Dose A); Sentinel Cohort: RSV/hMPV Group 1 (Dose A)
Biological: RSV/hMPV vaccine candidate Dose B — Pharmaceutical form:Suspension for injection-Route of administration:Intramuscular Injection
  Arms: Booster Cohort-RSV/hMPV; Main Cohort: RSV/hMPV Group 2 (Dose B); Sentinel Cohort: RSV/hMPV Group 2 (Dose B)
Biological: Placebo — Pharmaceutical form:Suspension for injection-Route of administration:Intramuscular Injection
  Arms: Booster Cohort-Placebo; Main Cohort: Placebo-Group 3; Sentinel Cohort: Placebo-Group 3

SUMMARY:
The purpose of this study is to assess the safety and immunogenicity of a single intramuscular (IM) injection of different doses of an respiratory syncytial virus (RSV) and human metapneumovirus (hMPV) vaccine candidate, in adult participants aged 60 years and older. In addition, the study will evaluate the safety and immunogenicity of a booster vaccination administered 12 months after the primary vaccination in a subset of the study population.

DETAILED DESCRIPTION:
Study duration per participant:

12 months for the Sentinel and Main Cohorts and 24 months overall for the subset of participants enrolled in the Booster Cohort.

Treatment Duration:

Sentinel Cohort: 1 IM injection. Participants will be followed for 12 months post-vaccination.

Main Cohort: 1 IM injection. Participants will be followed for 12 months post-vaccination.

Booster Cohort: 1 IM injection 12 months after the primary vaccination (Main Cohort). Participants will be followed for 12 months after administration of the booster dose.

ELIGIBILITY:
Inclusion Criteria:

* Aged 60 years or older on the day of inclusion
* A female participant is eligible to participate if she is not pregnant or breastfeeding and is of non-childbearing potential.
* Participants who are determined by medical history, physical examination (if required), and clinical judgment of the investigator to be eligible for inclusion Note: Participants with pre-existing stable disease, defined as disease not requiring significant change in therapy or hospitalization for worsening disease during the 6 weeks before enrollment, can be included.

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

* Any screening laboratory parameter with laboratory abnormalities deemed clinically significant by the investigator
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy. Persons living with stable human immunodeficiency virus (HIV) are not excluded
* Known systemic hypersensitivity to any of the study intervention components (eg, polyethylene glycol, polysorbate); history of a life-threatening reaction to the study interventions used in the study or to a product containing any of the same substances; any allergic reaction (eg, anaphylaxis) after administration of mRNA coronavirus disease 2019 (COVID-19) vaccine
* History of RSV and/or hMPV-associated illness, diagnosed clinically, serologically, or microbiologically in the last 12 months
* Previous history of myocarditis, pericarditis, and/or myopericarditis
* Screening electrocardiogram that is consistent with possible myocarditis, pericarditis, and/or myopericarditis or, in the opinion of the investigator, demonstrates clinically relevant abnormalities that may affect participant safety or study results
* Thrombocytopenia or bleeding disorder, contraindicating intramuscular (IM) injection based on investigator's judgment
* Receipt of anticoagulants in the 3 weeks preceding inclusion
* Chronic illness that, in the opinion of the investigator, is at a stage where it might interfere with study conduct or completion
* Alcohol, prescription drug, or substance abuse that, in the opinion of the investigator, might interfere with the study conduct or completion
* History of acute infection symptoms or a positive severe acute respiratory syndrome coronavirus reverse transcription polymerase chain reaction (SARS-CoV-2 RT-PCR) or antigen test in the 10 days prior to the visit. A prospective participant should not be included in the study until the condition has resolved
* Receipt of any vaccine other than mRNA vaccine in the 4 weeks preceding any study intervention administration or planned receipt of any vaccine other than mRNA vaccine in the 4 weeks following any study intervention administration
* Receipt of any mRNA vaccine in the 60 days preceding any study intervention administration or planned receipt of any mRNA vaccine in the 60 days following any study intervention administration
* Previous vaccination against RSV and/or hMPV (with a licensed or investigational vaccine either as a monovalent vaccine or any combination of the antigens)
* Receipt of immune globulins, blood, or blood-derived products in the past 3 months
* Participation at the time of study enrollment (or in the 4 weeks preceding the first study intervention administration) or planned participation during the present study period in another clinical study investigating a vaccine, drug, medical device, or medical procedure The above information is not intended to contain all considerations relevant to a potential participation in a clinical trial.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 646 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2026-03-10 (Estimated); Study Completion 2026-03-10 (Estimated)

PRIMARY OUTCOMES:
Presence of unsolicited systemic immediate adverse events (AEs) | Within 30 minutes after primary vaccination
  Number of participants experiencing immediate an immediate unsolicited systemic adverse event
Presence of solicited injection site or systemic reactions | Within 7 days after primary vaccination
  Number of participants reporting:
  * injection site reactions: pain, erythema and swelling
  * systemic reactions: fever, headache, fatigue, myalgia, arthralgia and chills
Presence of unsolicited AEs | Within 28 days after vaccination
  Number of participants experiencing unsolicited AEs
Presence of medically attended adverse events (MAAEs) | Up to 6 months after primary injection
  Number of participants experiencing MAAEs
Presence of serious adverse events (SAEs) | Up to 6 months after primary injection
  Number of participants experiencing SAEs
Presence of adverse events of special interest (AESIs) | Up to 6 months after primary injection
  Number of participants experiencing AESIs
Presence of related SAEs | Throughout study (approximately 24 months)
  Number of participants experiencing related SAEs
Presence of related AESIs | Throughout study (approximately 24 months)
  Number of participants experiencing related AESIs
Presence of fatal SAEs | Throughout study (approximately 24 months)
  Number of participants experiencing fatal SAEs
Presence of out-of-range biological test results | Within 7 days after vaccination
  Number of participants with biological safety assessment values out of normal range (as per the laboratory performing the test, including shift from baseline values)
RSV-A serum neutralizing antibody (nAb) titers at pre-vaccination (D01) and 28 days post- primary vaccination (D29) in Phase IIa (Main/Booster Cohort) | Day 1 and Day 29
  RSV-A serum neutralizing antibody (nAb) titers at pre-vaccination (D01) and 28 days post- primary vaccination (D29)
hMPV serum nAb titers at pre-vaccination (D01), 28 days post-primary vaccination (D29) in Phase IIa (Main/Booster Cohort) | Day 1 and Day 29
  hMPV serum nAb titers at pre-vaccination (D01), 28 days post-primary vaccination (D29)

SECONDARY OUTCOMES:
RSV-A serum neutralizing antibody (nAb) titers at pre-vaccination (D01) and 28 days post-primary vaccination (D29) | Day 1 and Day 29
  RSV-A serum nAb titers at pre-vaccination (D01), 28 days (D29) post-primary vaccination
RSV-B serum neutralizing antibody (nAb) titers at pre-vaccination (D01) and 28 days post-primary vaccination (D29) | Day 1 and Day 29
  RSV-B serum nAb titers at pre-vaccination (D01), 28 days (D29) post-primary vaccination
hMPV serum nAb titers at pre vaccination (D01), 28 days post-primary vaccination (D29) | Day 1 and Day 29
  hMPV serum nAb titers at pre-vaccination (D01), 28 days (D29) post-primary vaccination
RSV A serum nAb titers at pre-vaccination (D01), 28 days (D29), 3, 6, 9 and 12 months post-primary vaccination | Day 1, Day 29, Month 3, Month 6, Month 9 and Month 12
  RSV A serum nAb titers at pre-vaccination (D01), 28 days (D29), 3, 6, 9 and 12 months post-primary vaccination
RSV B serum nAb titers at pre-vaccination (D01), 28 days (D29), 3, 6, 9 and 12 months post-primary vaccination | Day 1, Day 29, Month 3, Month 6, Month 9 and Month 12
  RSV B serum nAb titers at pre-vaccination (D01), 28 days (D29), 3, 6, 9 and 12 months post-primary vaccination
RSV A serum anti-F immunoglobulin G (IgG) antibody (Ab) titers at pre-vaccination (D01), 28 days (D29), 3, 6, 9 and 12 months post-primary vaccination | Day 1, Day 29, Month 3, Month 6, Month 9 and Month 12
  RSV A serum anti-F immunoglobulin G (IgG) antibody (Ab) titers at pre-vaccination (D01), 28 days (D29), 3, 6, 9 and 12 months post-primary vaccination
hMPV A serum nAb titers at pre vaccination (D01), 28 days (D29), 3, 6, 9 and 12 months post-primary vaccination | Day 1, Day 29, Month 3, Month 6, Month 9 and Month 12
  hMPV A serum nAb titers at pre vaccination (D01), 28 days (D29), 3, 6, 9 and 12 months post-primary vaccination
hMPV A serum anti-F IgG Ab titers at pre vaccination (D01), 28 days (D29), 3, 6, 9 and 12 months post-primary vaccination | Day 1, Day 29, Month 3, Month 6, Month 9 and Month 12
  hMPV A serum anti-F IgG Ab titers at pre vaccination (D01), 28 days (D29), 3 months (D91), and 6 months (D181) post vaccination
RSV A serum nAb titers at pre booster vaccination (D01), 28 days (D29), and 3, 6, 9, and 12 months post-booster vaccination | Day 1, Day 29, Month 3, Month 6, Month 9 and Month 12
  RSV A serum nAb titers at pre booster vaccination (D01), 28 days (D29), and 3, 6, 9, and 12 months post-booster vaccination
RSV B serum nAb titers at pre booster vaccination (D01), 28 days (D29), and 3, 6, 9, and 12 months post-booster vaccination | Day 1, Day 29, Month 3, Month 6, Month 9 and Month 12
  RSV B serum nAb titers at pre booster vaccination (D01), 28 days (D29), and 3, 6, 9, and 12 months post-booster vaccination
RSV A serum anti-F IgG Ab titers at pre-booster vaccination (D01), 28 days (D29), and 3, 6, 9, and 12 months post- booster vaccination | Day 1, Day 29, Month 3, Month 6, Month 9 and Month 12
  RSV A serum anti-F IgG Ab titers at pre-booster vaccination (D01), 28 days (D29), and 3, 6, 9, and 12 months post- booster vaccination
hMPV A serum nAb titers at pre booster vaccination (D01), 28 days (D29), and 3, 6, 9, and 12 months post booster vaccination | Day 1, Day 29, Month 3, Month 6, Month 9 and Month 12
  hMPV A serum nAb titers at pre booster vaccination (D01), 28 days (D29), and 3, 6, 9, and 12 months post-booster vaccination
hMPV serum anti-F IgG Ab titers at pre booster vaccination (D01), 28 days (D29), and 3, 6, 9, and 12 months post booster vaccination | Day 1, Day 29, Month 3, Month 6, Month 9 and Month 12
  hMPV serum anti-F IgG Ab titers at pre booster vaccination (D01), 28 days (D29), and 3, 6, 9, and 12 months post- booster vaccination

CONTACTS AND LOCATIONS:
Locations (13):
- United States (10):
  - Collaborative Neuroscience Research Site Number : 8400017, Los Alamitos, California
  - Matrix Clinical Research Site Number : 8400011, Los Angeles, California
  - Peninsula Research Associates Site Number : 8400001, Rolling Hills Estates, California
  - Suncoast Research Associates, LLC Site Number : 8400002, Miami, Florida
  - AMR Chicago, Oakbrook Terrace Site Number : 8400019, Oakbrook Terrace, Illinois
  - Velocity Clinical Research, Sioux City Site Number : 8400012, Sioux City, Iowa
  - AMR Lexington Site Number : 8400008, Lexington, Kentucky
  - AMR Kansas City Site Number : 8400014, Kansas City, Missouri
  - AMR Knoxville Site Number : 8400010, Knoxville, Tennessee
  - DM Clinical Research - Tomball Site Number : 8400004, Tomball, Texas
- Puerto Rico (3):
  - Investigational Site Number : 6300002, Guayama
  - Investigational Site Number : 6300001, San Juan
  - Investigational Site Number : 6300003, San Juan

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: VBD00003 Plain Language Results Summaries — https://www.trialsummaries.com/Study/StudyDetails?id=25526&tenant=MT_SNY_9011